CLINICAL TRIAL: NCT02720458
Title: Self-help Program for Hypnotics Withdrawal in Chronic Insomniac Patients: A Randomized Controlled Clinical Trial
Brief Title: Self Help Program for Hypnotics Withdrawal in Insomniac Patients
Acronym: PROPERSOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX 2014/35
Record Dates: First submitted 2016-03-10; First posted 2016-03-28 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Insomnia
Keywords: Hypnotics withdrawal in insomniac patients; Cognitive-Behavioural Therapy (CBT); Internet-delivered self-help program; Sleep restriction; Stimulus control; Half-life benzodiazepine; Z-drug
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standardized hypnotic taper and self-help program (Experimental)
  Interventions: Other: Standardized gradual hypnotic taper; Behavioral: Short-term simple self-help program
- Standardized hypnotic taper only (Active Comparator)
  Interventions: Other: Standardized gradual hypnotic taper

INTERVENTIONS:
Other: Standardized gradual hypnotic taper — The gradual hypnotic taper is standardized and is adjusted depending on the hypnotic treatment and the initial weekly dose. The practitioner will give to the patient a calendar for the taper period with the specific dose for each day (name of hypnotic, quantity and dose of pills).
Behavioral: Short-term simple self-help program — The short-term simple self-help program consists in:
  * Restriction of time in bed
  * Stimulus control instructions
  The restriction of time in bed would be delivered by an e-health tool (web site). The patient will have to connect to the web site with an individual connexion password. He will connect every day to complete an on-line sleep diary during the period of the simple short-term behavioural program (5 weeks). After this period, patients will have the choice to continue connecting to the website and using the program or to stop using the program.
  Arms: Standardized hypnotic taper and self-help program

SUMMARY:
Persistent insomnia has a high prevalence in French general population affecting between 15.8 % and 19 % of adults. In France, the disease is mainly managed by general practitioners (GP) who usually proposed intermediate half-life benzodiazepines and Z-drugs in first-line treatment. French Health authorities recommend restricting the consumption of both hypnotics to no more than 4 weeks, considering their potential adverse effects (memory impairment, altered sleep physiology, motor-vehicle crash), and the risk of tolerance and dependence. However, it appears that a majority of patients become chronic users. Therefore, discontinuation of benzodiazepines/Z-drugs is recommended, but it may appear as a challenge due to withdrawal symptoms and psychological factors (anticipatory anxiety, fear of rebound insomnia).

Numerous studies have shown that programs based on Cognitive-Behavioural Therapy (CBT) principles improve sleep and daily life quality leading to hypnotic taper and maintain of hypnotic abstinence in insomniac patients. Cognitive-Behavioural Therapy (CBT) is based on 4 components: sleep restriction, stimulus control, cognitive therapy and sleep hygiene education. This therapy is dependent on a therapeutic alliance between practitioner and patient. Unfortunately, there are an insufficient number of trained CBT experts especially in France.

The implementation of an internet-delivered self-help program based on time-in-bed restriction and stimulus control may be an issue within the context of general practice.

Online programs based on CBT principles have been proved to be effective in improving the sleep and daytime functioning in this population, but the studies were realized in small patients groups.

Investigators hypothesis is that a simple and internet-delivered short-term program based on sleep restriction therapy and stimulus control (following to a GP consultation) may facilitate hypnotics discontinuation (benzodiazepines/Z-drugs) in patient with insomnia disorder still reporting sleep complaints in comparison with a tapering alone (no access to the self-help program).

ELIGIBILITY:
Inclusion Criteria:

* Patient complaining of persistent insomnia without co-morbidities (DSM-5) and treated for at least 3 months with monotherapy of:
* Zopiclone or Zolpidem with usual doses (3.5 doses per week at least to a maximum of 14 per week) OR Intermediate half-life benzodiazepines included in the appendix 1 list with usual doses (3.5 doses per week at least to a maximum of 14 per week)
* Motivated to stop hypnotic treatment (score >5 on a 1 to 10 degrees VAS)
* 18 to 75 years old,
* Man or woman,
* Having an internet connection,
* Affiliated to a national health service,
* Having given written informed consent to participate in the trial.

Exclusion Criteria:

* Patient with 2 psychotropic drugs or more taken daily for insomnia complaints (antidepressant, anxiolytic and antihistamine treatments will be allowed if they are prescribed for a stabilized mood and/or anxiety disorder).
* Patient not believing in short-term simple self-help program
* Insomnia with comorbidities other than a stabilized mood and/or anxiety disorder
* Night and shift-workers,
* Current Psychiatric disorder : mood disorder (depression, bipolar disorder) with a BDI score > 19, anxiety disorder, psychosis
* All sleep disorders other than persistent insomnia (clinical interview),
* Progressive neurological diseases that include restless legs syndrome,
* Unstable Cardiovascular disease,
* Unstable respiratory or endocrinological diseases (clinical interview),
* Drug addiction, alcohol addiction during the previous 6 months (clinical interview),
* Having undertaken trans-meridian travel (± 3H) in the previous 1 month
* Pregnant or lactating woman,
* Current participation in psychotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Urinary hypnotics screening assessed during Visit 2 | 7 weeks after randomization visit
  Urine will be frozen and afterwards analysed by a central laboratory (Unité de biologie médicale multidisciplinaire, CHU Bordeaux) for hypnotics (benzodiazepines and Z-drugs) using Gas Chromatography-Mass Spectrometry.

SECONDARY OUTCOMES:
Urinary hypnotics screening assessed during Visit 3 | 17 weeks after randomization visit
  Urine will be frozen and afterwards analysed by a central laboratory (Unité de biologie médicale multidisciplinaire, CHU Bordeaux) for hypnotics (benzodiazepines and Z-drugs) using Gas Chromatography-Mass Spectrometry.
Total sleep time obtained by actimetry | During 10 nights before Visit 2 wich is scheduled 7 weeks after randomization visit
Sleep efficiency obtained by actimetry | During 10 nights before Visit 2 wich is scheduled 7 weeks after randomization visit
Wake after sleep onset obtained by actimetry | During 10 nights before Visit 2 wich is scheduled 7 weeks after randomization visit
Sleep latency obtained by actimetry | During 10 nights before Visit 2 wich is scheduled 7 weeks after randomization visit
Total sleep time obtained by sleep diary | Every night between Pre-Inclusion visit (Visit 0) and Week 5 after Visit 1
Sleep efficiency obtained by sleep diary | Every night between Pre-Inclusion visit (Visit 0) and Week 5 after Visit 1
Wake after sleep onset obtained by sleep diary | Every night between Pre-Inclusion visit (Visit 0) and Week 5 after Visit 1
Sleep latency obtained by sleep diary | Every night between Pre-Inclusion visit (Visit 0) and Week 5 after Visit 1
Insomnia Severity Scale (ISI) score | Pre-inclusion visit (between 21 to 10 days before randomization), randomization visit (Visit 1) ,7 weeks after randomization (Visit 2) and 17 weeks after randomization (Visit 3)
Leeds Sleep Evaluation Questionnaire (LSEQ) score | 7 weeks after randomization (Visit 2) and 17 weeks after randomization (Visit 3)
Beck Depression Inventory Second Edition (BDI-II) score | Pre-inclusion visit (between 21 to 10 days before randomization), randomization visit (Visit 1) ,7 weeks after randomization (Visit 2) and 17 weeks after randomization (Visit 3)
Beck anxiety Inventory (BAI) score | Pre-inclusion visit (between 21 to 10 days before randomization), randomization visit (Visit 1) ,7 weeks after randomization (Visit 2) and 17 weeks after randomization (Visit 3)
Short-Form SF-36 Health Survey score | Pre-inclusion visit (between 21 to 10 days before randomization), randomization visit (Visit 1) ,7 weeks after randomization (Visit 2) and 17 weeks after randomization (Visit 3)
Benzodiazepine Withdrawal Symptoms Questionnaire (BWSQ) score | 7 weeks after randomization (Visit 2) and 17 weeks after randomization (Visit 3)
Self-efficiency visual analog scale score | Pre-inclusion visit (between 21 to 10 days before randomization), randomization visit (Visit 1) and 7 weeks after randomization (Visit 2)
Reasons for non-compliance obtained during patient interview | 7 weeks after randomization (Visit 2) and 17 weeks after randomization (Visit 3)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine BENARD, MD-PhD, Study Chair — USMR - CHU de Bordeaux
Locations (6):
- France (6):
  - CHU de Bordeaux, Bordeaux
  - APHP Hôpital Raymond Poincaré, Garches
  - CHRU de Lille, Lille
  - CHU de Montpellier, Montpellier
  - AP-HP Hôpital Pitié-Salpétrière, Paris
  - APHP Hôtel-Dieu de Paris, Paris

IPD SHARING:
Plan to Share IPD: Yes
Patient could request investigator an access to IPD according to French regulation (act No. 78-17 of 6 January 1978 on data processing, data files and individual liberties, amended by act No. 2004-801 of 6 August 2004).